CLINICAL TRIAL: NCT00887003
Title: Effects of Volume and Dose of Local Anaesthetic Solution in Epidural Steroidal Injections for Patients With Chronic Lower Back Pain
Brief Title: Epidural Study of Patients With Chronic Lower Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 04-392
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Low Back Pain
Keywords: epidural; volume; dose; pain relief; steroid
MeSH Terms: interventions — Bupivacaine; Steroids; Methylprednisolone Acetate; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LV/LD 1 (Experimental): Low Volume, Low Dose (5cc, 5mg plain Bupivacaine) + 80mg Depo-Medrol
  Interventions: Drug: Bupivacaine; Drug: Depo-Medrol
- LV/HD 2 (Experimental): Low Volume, High Dose (5cc, 10mg plain Bupivacaine) + 80mg Depo-Medrol
  Interventions: Drug: Bupivacaine; Drug: Depo-Medrol
- HV/LD 3 (Experimental): High Volume, Low Dose (10cc, 5mg plain Bupivacaine) + 80mg Depo-Medrol
  Interventions: Drug: Bupivacaine; Drug: Depo-Medrol
- HV/HD 4 (Experimental): High Volume, High Dose (10cc, 10mg plain Bupivacaine) + 80mg Depo-Medrol
  Interventions: Drug: Bupivacaine; Drug: Depo-Medrol

INTERVENTIONS:
Drug: Bupivacaine — Low Volume, Low Dose (5cc, 5mg plain Bupivacaine)
  Other Names: steroid
  Arms: LV/LD 1
Drug: Bupivacaine — Low Volume, High Dose (5cc, 10mg plain Bupivacaine)
  Other Names: steroid
  Arms: LV/HD 2
Drug: Bupivacaine — High Volume, Low Dose (10cc, 5mg plain Bupivacaine)
  Other Names: steroid
  Arms: HV/LD 3
Drug: Bupivacaine — High Volume, High Dose (10cc, 10mg plain Bupivacaine)
  Other Names: steroid
  Arms: HV/HD 4
Drug: Depo-Medrol — 80mg Depo-Medrol
  Other Names: methylprednisolone

SUMMARY:
The purpose of this study is to examine 4 different epidural dosing regimes of local anaesthetic solution in a series of 3 epidural injections over a period of 12 months to determine the optimum dose of anaesthetic solution for pain relief and to determine the nature of any adverse events by measuring anxiety and depression, functionality and any side effects of the medication.

DETAILED DESCRIPTION:
To determine the optimum dose of local anesthetic and the optimum volume of injected solution when used in an epidural steroid injection being given for pain relief to patients with chronic lower back pain, using pain scores as an assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* lower back pains > 6 months
* no lumbar epidural in past 6 months
* no previous back surgery
* written informed consent to participate in study

Exclusion Criteria:

* acute lower back pain
* pregnancy
* significant psychiatric disease
* local or systemic infection
* coagulopathy/anticoagulant therapy
* bleeding diathesis
* presently enrolled in another study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2005-05; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The volume and dose of local anesthetic injected epidurally, in combination with the steroid, will be measured against the duration and degree of pain relief. | Pain scores will be measured at 6 time intervals throughout the study period, prior to 1st injection, 30 minutes post 1st injection, prior to 2nd injection and 3rd injections and at 3 and 6 month post the three month injection.

SECONDARY OUTCOMES:
Secondary outcomes will be scores on the Oswestry low back pain disability scale and the Hospital anxiety and depression scale correlated with treatment outcomes and adverse events. | Oswestry scores and HADS scores will be calculated at 5 time periods throughout the study period, prior to 1st, 2nd, and 3rd injections and at 3 and 6 month post the three month injection.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Mulcaster, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada